CLINICAL TRIAL: NCT04961294
Title: Electrical Acupuncture for Protracted Withdrawal of Opioid Use Disorder: A Pragmatic Randomized Controlled Trial
Brief Title: EA for Protracted Withdrawal of OUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ren Yu-Lan, professor, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018SZ071
Record Dates: First submitted 2021-05-26; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-Acupuncture group (Experimental): The patients in this group will be treated with electro-acupuncture for 30 minutes twice a week in a month. We conduct Nei Guan (PC6), Shen Men (HT7), ZuSanli (ST36), SanYinjiao (SP6) as the major points. Each time treating, according to other symptoms, we will give no more than 2 additional points.
  Interventions: Device: Electro-Acupuncture
- Wait-list group (No Intervention): We give no intervention to the patients this group during the whole experiment. When finishing, the same ways of treatment will be given to these patients.

INTERVENTIONS:
Device: Electro-Acupuncture — Acupuncture used for thousands years is part of traditional Chinese medicine. We use electro-acupuncture to treat our patients because it is more sufficient than traditional acupuncture and proved effectively treating protracted withdrawal syndrome of opioid use disorder. Paired alligator clips of the EA apparatus will be attached to the needle holders of Shenmen and Neiguan points on both sides. EA stimulation will last for 30 min with a continuous wave of 2/100Hz and intensity of 10-15 mA which patients can stand. All needles will be removed in 30 min and use a dry sterilised cotton ball to press the points in case of bleeding.
  Arms: Electro-Acupuncture group

SUMMARY:
Opioid use disorder (OUD) the most harmful of all the illicit drugs is a serious substance-related disorder resulting from abuse or misuse of opioids. Huge number of patients are addictive to opioid and evidences show that patients with OUD have high rates of infectious diseases.The "World Drug Report 2020" has declared that 58 million people used opioids in 2018 and some 35.6 million people suffered from drug use disorders globally. More than 11 million people inject drugs, while 1.4 million PWID are living with HIV, 5.5 million with hepatitis C and 1.2 million are living with both hepatitis C and HIV.

The long-term physical and mental symptoms of some opioid drug users after detoxification treatment are called protracted opioid withdrawal syndrome (POAS). POAS is one of the important causes of relapse. Methadone maintenance treatment is the most widespread and extensively researched treatment for heroin addiction and has been shown to reduce the frequency of opioid use, the mortality, and the transmission of human immunodeficiency virus and viral hepatitis. But higher daily methadone dose and increasing duration of treatment conduce the addiction in methadone. Other medication therapy like naltrexone treatment is also associated with high rates of noncompliance and opioid relapse. Meanwhile, relapse to heroin use following cessation of agonist maintenance treatment is common. The problems associated with use of opioid agonists have made it necessary to develop non-opioid therapies to ameliorate the symptoms of acute and protracted opioid withdrawal.

Acupuncture based on traditional Chinese medicine (TCM) theory is becoming a popular complementary and alternative treatment worldwide. Study showed that acupuncture reduced the depression symptoms and cravings of patients under methadone maintenance treatment. Another study by Le et al. (2016) showed that electric acupuncture has been associated with a reduction in depressive symptoms through the adjustment of HPA axis function and increasing the hippocampus activity. And also some research show the efficiency of acupuncture in treating mice with OUD.

Investigators conduct a pragmatic randomized controlled trials(pRCT) to observe the effect of acupuncture in a larger sample. It combines the advantages of randomization and real-world data, and the results can provide the best real-world evidence for the assessment of intervention effects or comparative effects.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria
* the results of detection of morphine in urine is negative
* the patients must be conscious, with no aphasia, no intellectual disability, and graduate from primary school so they can understand what the scale mean and cooperate the treatment.
* not involved in any clinical trials in 3 months
* sign the Informed Consent Form

Exclusion Criteria:

* with any injury or infection around the acupoint
* the patients are intolerant or allergic to acupuncture or electro-acupuncture
* the women is pregnant or lactating
* patients whose heart, liver or kidney with severe impairment
* according to the judgement from investigators, patients don't correspond with this research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Opiate Withdrawal Syndrome Scale | Change from baseline Opiate Withdrawal Syndrome Scale scores at 1 month.
  It consists of three subscales, namely, "anxiety and mood", "fatigue", and "craving". Items are scored on a five-point scale ranging from 0 to 4 with higher scores representing more severe PAAS.

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAMD) | Change from baseline Hamilton Depression Scale scores at 1 month.
  Assessment for depression.And the interpretation of HAMD scores is as follows: <7, no depression; 7-17, mild depression; 17-24, moderate depression; and >24, severe depression.
Hamilton Anxiety Scale (HAMA) | Change from baseline Hamilton Anxiety Scale scores at 1 month.
  Assessment for anxiety. And the interpretation of HAMA scores is as follows: <7, no anxiety;7-14, mild anxiety; 14-20, moderate anxiety; 21-28, severe anxiety; and >29, extremely severe anxiety.
Pittsburgh sleep quality index (PSQI) | Change from baseline Pittsburgh sleep quality index scores at 1 month.
  The scores are from 0 to 21.Higher scores reflect worse sleep quality.
Concise health survey questionnaire | Change from baseline Concise health survey questionnaire scores at 1 month.All scores were recoded with 0 as a minimum score and 100 as a maximum score; a higher score indicates a better quality of life.
  This questionnaire contains 9 parts: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health and Reported Health Transition.
Dopamine (DA) | baseline and one month
  The physiological parameter to observe the efficiency of acupuncture.
5-hydroxytryptamine (5-HT) | Change from baseline 5-hydroxytryptamine at 1 month.
  The physiological parameter to observe the efficiency of acupuncture.
Liver function | Change from baseline alanine aminotransferase, aspartate aminotransferase, bilirubin total and direct bilirubin at 1 month.
  The physiological parameter to prove the safety of acupuncture.
Renal function | Change from baseline serum creatinine, blood uric acid and blood urea nitrogen at 1 month.
  The physiological parameter to prove the safety of acupuncture.
Testosterone | Change from baseline Testosterone at 1 month.
  The physiological parameter to observe the efficiency of acupuncture.
Prolactin (PRL) | Change from baseline Prolactin at 1 month.
  The physiological parameter to observe the efficiency of acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Yulan Ren, PhD, Study Chair — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Affliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China